CLINICAL TRIAL: NCT04318990
Title: Distal vs. Proximal Radial Artery Access for Cardiac Catheterization and Intervention
Brief Title: DIstal vs Proximal Radial Artery Access for Cath
Acronym: DIPRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 019-504 DIPRA
Record Dates: First submitted 2020-03-19; First posted 2020-03-24 (Actual); Results first posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2020-03

CONDITIONS: Coronary Angiography; Coronary Angioplasty

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, single-center clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Distal radial artery access (Experimental): Wrist rests on a comfortable underground which brings the wrist in passive ulnar flexion. Patient is asked to bring the thumb under the other four fingers. After disinfection, patient is covered with a sterile drape. Brachial drape is applied to the hand exposing the anatomical snuff box and the proximal radial. Under ultrasound guidance, local anesthesia applied by SC injection of 5cc of lidocaine filling the radial fossa. Puncture performed at the point of maximal pulsation proximal in the anatomical snuffbox. If fails, a puncture more distal, can be attempted. After successful anterior wall puncture a radial sheath wire is advanced. Proper position verified by fluoroscopy or by ultrasound to ensure the wire didn't traverse the palmar arch, followed by introduction of a hydrophilic sheath. After administration of a spasmolytic cocktail containing 200-400 mcg of nitroglycerin and 5 mg of verapamil, the operator can take up a position at the level of the patient's knees.
  Interventions: Procedure: Distal radial artery access
- Proximal radial artery access (Active Comparator): Half of the patients enrolled in the study undergoing coronary angiography or angioplasty at The Heart Hospital Baylor Plano will be randomized proximal radial access for cardiac catheterization.
  Interventions: Procedure: Proximal radial artery surgery

INTERVENTIONS:
Procedure: Distal radial artery access — Patients undergoing coronary angiography or angioplasty at The Heart Hospital Baylor Plano will be randomized 1:1 to distal or proximal radial access for cardiac catheterization.
  Arms: Distal radial artery access
Procedure: Proximal radial artery surgery — Patients undergoing coronary angiography or angioplasty at The Heart Hospital Baylor Plano will be randomized 1:1 to distal or proximal radial access for cardiac catheterization.
  Arms: Proximal radial artery access

SUMMARY:
This single-center, prospective, randomized study will evaluate distal radial artery (dRA) vs. proximal radial artery access (pRA) in regards to hand function and radial artery occlusion.

DETAILED DESCRIPTION:
Primary objective is to evaluate hand function following distal radial artery access compared to proximal artery access in patients undergoing cardiac catheterization.

Hand function will be assessed by:

* QuickDASH questionnaire
* Hand grip test
* Thumb forefinger pinch test utilizing a pinch gauge

Secondary objectives: Vascular access success rates, hematoma, bleeding, complications of vascular access and radial artery occlusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. The distal and proximal radial artery must be palpable and non-occlusive flow must be confirmed by (Doppler) ultrasound.
3. Patient should be able to comply with the protocol.
4. Provide written informed consent before study participation

Exclusion Criteria:

1. Obligatory femoral or forearm radial access
2. Previous ipsilateral forearm radial artery occlusion.
3. Patient on therapeutic oral anticoagulation.
4. Very large hand/wrist anatomy that will preclude using the available hemostatic radial bands.
5. Enrolment in another study that competes or interferes with this study.
6. Poor clinical condition like cardiogenic shock, which prohibits pre- and post-procedural function tests.
7. Subject with planned complex PCI or procedure necessitating multiple intervention.
8. Any other condition or co-morbidity which, in the opinion of the investigator or operator, may pose a significant hazard to the subject if he or she is enrolled in the study.
9. History of stroke with residual deficit that affects hand function.
10. Previous radial artery catheterization within 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor Scott & White The Heart Hospital - Plano, Plano, Texas, United States

REFERENCES:
- [Derived] Al-Azizi K, Moubarak G, Dib C, Sayfo S, Szerlip M, Thomas S, McCracken J, Smith A, Kelavkar U, Hale S, Van Zyl J, McCoy SL, Lanfear AT, Banwait JK, Ravindranathan P, Chionh K, DiMaio JM, Mack MJ, Potluri S. Distal Versus Proximal Radial Artery Access for Cardiac Catheterization: 30-Day Outcomes of the DIPRA Study. J Am Heart Assoc. 2023 Nov 7;12(21):e030774. doi: 10.1161/JAHA.123.030774. Epub 2023 Oct 27. PMID 37889176
- [Derived] Flumignan RL, Trevisani VF, Lopes RD, Baptista-Silva JC, Flumignan CD, Nakano LC. Ultrasound guidance for arterial (other than femoral) catheterisation in adults. Cochrane Database Syst Rev. 2021 Oct 12;10(10):CD013585. doi: 10.1002/14651858.CD013585.pub2. PMID 34637140

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who were undergoing a cardiac catheterization at Baylor Scott and White- The Heart Hospital Plano were considered for enrollment in the trial. Enrollment started in March 2020 and completed in December 2021.
Pre-assignment Details: Subjects who met the screening inclusion criteria and have not met any of the trial exclusion criteria were included in the study. Screening assessments were conducted through review of medical records and by interview after informed consent was signed. In addition, a mandatory screening assessment for research purposes included assessing the patency of the pRA and dRA using palpation first, and if both are palpable then doppler ultrasound.
Period: Overall Study
Arm/Group | Distal Radial Artery Access | Proximal Radial Artery Access
Started | 150 | 150
Completed | 112 | 104
Not Completed | 38 | 46

BASELINE CHARACTERISTICS:
Population: All patients enrolled and randomized in the DIPRA trial
Groups:
- Total: Total of all reporting groups
Arm/Group | Distal Radial Artery Access | Proximal Radial Artery Access | Total
Number analyzed (Participants) | 150 | 150 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (8.7) | 67.3 (10.5) | 66.6 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 43 | 74
  Male | 119 | 107 | 226
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 147 | 143 | 290
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 8 | 5 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 9 | 17
  White | 128 | 132 | 260
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 5 | 3 | 8
BMI [Mean (Inter-Quartile Range); unit: kg/m2] | 29.9 [26.8 to 34.1] | 30.1 [26.9 to 35.0] | 30.0 [26.8 to 34.4]
Diabetes Mellitus [Count of Participants; unit: Participants] | 51 | 45 | 96
Hypercholesteremia [Count of Participants; unit: Participants] | 27 | 29 | 56
Hypertension [Count of Participants; unit: Participants] | 112 | 120 | 232
Prior Myocardial Infarction [Count of Participants; unit: Participants] | 23 | 16 | 39
Prior CABG [Count of Participants; unit: Participants] | 3 | 3 | 6
Prior PCI [Count of Participants; unit: Participants] | 25 | 31 | 56

OUTCOME MEASURES:

1. Primary Outcome: Quick Disabilities of the Arm Shoulder and Hand (DASH) Questionnaire Score (0-100)
Description: Hand function questionnaire, Range: 0 (no disability) to 100 (most severe disability)
Time Frame: 1 year
Population: Patients who completed 1 year of follow up
Measure: Median (Inter-Quartile Range); unit: DASH Score change from baseline
Arm/Group | Distal Radial Artery Access | Proximal Radial Artery Access
Number analyzed (Participants) | 112 | 104
DASH Score change from baseline | 0 [-6.6 to 2.3] | 0 [-4.6 to 2.9]

2. Primary Outcome: Thumb and Forefinger Pinch Strength Test
Description: Hand function: Thumb and forefinger pinch strength (kg)
Time Frame: 1 year
Population: Patients who completed 1 year of follow up
Measure: Median (Inter-Quartile Range); unit: pinch grip(kg) change from baseline
Arm/Group | Distal Radial Artery Access | Proximal Radial Artery Access
Number analyzed (Participants) | 112 | 104
pinch grip(kg) change from baseline | -0.1 [-1.1 to 1] | -0.3 [-1 to 0.7]

3. Primary Outcome: Hand Grip Strength Test
Description: Hand grip strength test (kg)
Time Frame: 1 month
Population: Patients who completed 1 year of follow up
Measure: Median (Inter-Quartile Range); unit: hand grip (kg) change from baseline
Arm/Group | Distal Radial Artery Access | Proximal Radial Artery Access
Number analyzed (Participants) | 112 | 104
hand grip (kg) change from baseline | 0.7 [-3 to 4.5] | 1.3 [-2 to 4.3]

4. Secondary Outcome: Re-intervention Using the Radial Artery
Description: Patients who required re-intervention using the radial artery up to 1 year following the initial intervention
Time Frame: 1 year
Population: Patients who completed 1 year of follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Distal Radial Artery Access | Proximal Radial Artery Access
Number analyzed (Participants) | 112 | 104
Participants | 5 | 8

5. Secondary Outcome: Radial Artery Occlusion
Description: Occurrence of distal radial artery occlusion and proximal radial artery occlusion for patients who had distal or proximal radial artery access
Time Frame: 1 year
Population: Patients who completed 1 year of follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Distal Radial Artery Access | Proximal Radial Artery Access
Number analyzed (Participants) | 112 | 104
Participants
  Distal | 0 | 2
  Proximal | 0 | 1
  No Radial Artery Occlusion | 112 | 101

ADVERSE EVENTS:
Time Frame: 1 year
Description: The adverse events monitored until 1 year after the index procedure are complications to related to the procedure including bleeding, hematoma, and radial occlusion. Serious adverse events are defined as usual, but exclude hospitalizations for treatment, which was elective or preplanned, for a pre-existing condition unrelated to the study and did not worsen and for outpatient emergency treatment for an event not fulfilling any of the definitions of serious not resulting in hospital admission.
Arm/Group | Distal Radial Artery Access | Proximal Radial Artery Access
All-Cause Mortality (participants affected / at risk) | 1/150 | 1/150
Serious Adverse Events (participants affected / at risk) | 4/150 | 1/150
Other Adverse Events (participants affected / at risk) | 0/150 | 0/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Distal Radial Artery Access (N=150) | Proximal Radial Artery Access (N=150)
Acute respiratory failure with hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Orthopedic Injury (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Gross hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-24): https://cdn.clinicaltrials.gov/large-docs/90/NCT04318990/Prot_SAP_000.pdf
  • Informed Consent Form (2020-02-05): https://cdn.clinicaltrials.gov/large-docs/90/NCT04318990/ICF_001.pdf